CLINICAL TRIAL: NCT01640002
Title: A Randomized, Placebo-Controlled Study to Assess the Efficacy of Propantheline for the Treatment of Overactive Bladder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Jose Abraao Carneiro Neto, MD, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FR-473218
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Overactive Bladder Associated With HTLV-1
Keywords: overactive bladder; HTLV-1; Propantheline; anticholinergic
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Propantheline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propantheline (Active Comparator)
  Interventions: Drug: Propantheline Bromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propantheline Bromide — 15MG OF PROPANTHELINE BROMIDE, THREE TIMES DAILY FOR 02 MONTHS.
  Arms: Propantheline
Drug: Placebo — PLACEBO CAPSULE, 03 TIMES DAILY FOR 02 MONTHS
  Arms: Placebo

SUMMARY:
It's a double blind, placebo controlled study to assess the efficacy of Propantheline Bromide to treat overactive bladder (OAB) in HTLV 1 infected patients.

We think that the treatment of the OAB with Propantheline could reduce nocturia and frequency in sixty percent.

DETAILED DESCRIPTION:
Double blind, placebo controlled study to assess the efficacy of Propantheline Bromide to treat overactive bladder (OAB) in HTLV 1 infected patients

Treatment Group Propantheline Bromide: 15mg, three times daily for 08 weeks.

Control Group Placebo 03 times daily

Case definition Clinically defined OAB patients (ICS criteria), infected by HTLV-1. Frequency was defined as more than 08 daytime voids. Nocturia was defined as more than 02 voids after sleeping.

Inclusion criteria More than 18 year. HTLV-1 infected patients with overactive bladder. Negative culture of urine. Without neurological impairment.

Exclusion criteria Persistently positive urine culture

History of:

Allergy to medication, head or spinal trauma. Head and neck, neurological,spinal, lower abdominal or pelvic surgery. Stroke. Users of urinary catheters.

ELIGIBILITY:
Inclusion Criteria:

* HTLV-1 infection
* More than 18 years
* Negative urine culture
* No neurological damage

Exclusion Criteria:

* Diabetes
* Persistently positive urine culture
* Pelvic, head, urological or gynecological surgery
* Stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Improve in Overactive bladder symptoms score | 2 months

SECONDARY OUTCOMES:
Improvement in nocturia and urgency | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: José Abraão Carneiro Neto, Principal Investigator — Service of Imunology - Universitary Hospital Prof. Edgard Santos
Locations (1):
- Service of Imunology - Universitary Hospital Prof. Edgard Santos, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Rocha PN, Rehem AP, Santana JF, Castro N, Muniz AL, Salgado K, Rocha H, Carvalho EM. The cause of urinary symptoms among Human T Lymphotropic Virus Type I (HLTV-I) infected patients: a cross sectional study. BMC Infect Dis. 2007 Mar 12;7:15. doi: 10.1186/1471-2334-7-15. PMID 17352816
- [Background] Poetker SK, Porto AF, Giozza SP, Muniz AL, Caskey MF, Carvalho EM, Glesby MJ. Clinical manifestations in individuals with recent diagnosis of HTLV type I infection. J Clin Virol. 2011 May;51(1):54-8. doi: 10.1016/j.jcv.2011.02.004. Epub 2011 Mar 8. PMID 21388871
- [Background] Caskey MF, Morgan DJ, Porto AF, Giozza SP, Muniz AL, Orge GO, Travassos MJ, Barron Y, Carvalho EM, Glesby MJ. Clinical manifestations associated with HTLV type I infection: a cross-sectional study. AIDS Res Hum Retroviruses. 2007 Mar;23(3):365-71. doi: 10.1089/aid.2006.0140. PMID 17411369
- [Background] Gomes I, Melo A, Proietti FA, Moreno-Carvalho O, Loures LA, Dazza MC, Said G, Larouze B, Galvao-Castro B. Human T lymphotropic virus type I (HTLV-I) infection in neurological patients in Salvador, Bahia, Brazil. J Neurol Sci. 1999 May 1;165(1):84-9. doi: 10.1016/s0022-510x(99)00083-0. PMID 10426153
- [Background] Garlet GP, Giozza SP, Silveira EM, Claudino M, Santos SB, Avila-Campos MJ, Martins W Jr, Cardoso CR, Trombone AP, Campanelli AP, Carvalho EM, Silva JS. Association of human T lymphotropic virus 1 amplification of periodontitis severity with altered cytokine expression in response to a standard periodontopathogen infection. Clin Infect Dis. 2010 Feb 1;50(3):e11-8. doi: 10.1086/649871. PMID 20038241
- [Background] Tannus M, Tanajura D, Sundberg MA, Oliveira P, Castro N, Santos AM. Detrusor Arreflexia as an End Stage of Neurogenic Bladder in HAM/TSP? Case Rep Med. 2011;2011:289389. doi: 10.1155/2011/289389. Epub 2011 Apr 13. PMID 21541226
- [Background] Thuroff JW, Bunke B, Ebner A, Faber P, de Geeter P, Hannappel J, Heidler H, Madersbacher H, Melchior H, Schafer W, et al. Randomized, double-blind, multicenter trial on treatment of frequency, urgency and incontinence related to detrusor hyperactivity: oxybutynin versus propantheline versus placebo. J Urol. 1991 Apr;145(4):813-6; discussion 816-7. doi: 10.1016/s0022-5347(17)38459-8. PMID 2005707
- [Background] Gotoh M, Homma Y, Yokoyama O, Nishizawa O. Responsiveness and minimal clinically important change in overactive bladder symptom score. Urology. 2011 Oct;78(4):768-73. doi: 10.1016/j.urology.2011.06.020. PMID 21855969
- [Result] Castro NM, Rodrigues W Jr, Freitas DM, Muniz A, Oliveira P, Carvalho EM. Urinary symptoms associated with human T-cell lymphotropic virus type I infection: evidence of urinary manifestations in large group of HTLV-I carriers. Urology. 2007 May;69(5):813-8. doi: 10.1016/j.urology.2007.01.052. PMID 17482910
- [Result] Oliveira P, Castro NM, Muniz AL, Tanajura D, Brandao JC, Porto AF, Carvalho EM. Prevalence of erectile dysfunction in HTLV-1-infected patients and its association with overactive bladder. Urology. 2010 May;75(5):1100-3. doi: 10.1016/j.urology.2009.11.041. Epub 2010 Feb 26. PMID 20189229